CLINICAL TRIAL: NCT02194374
Title: A Study to Infuse ROR1-Specific Autologous T Cells for Patients With Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
Brief Title: Autologous ROR1R-CAR-T Cells for Chronic Lymphocytic Leukemia (CLL)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed with no enrollment due to unavailability of reagent.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CLL Global Research Foundation Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0932; NCI-2014-01715 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic lymphocytic leukemia; CLL; Small lymphocytic lymphoma; SLL; B cell; ROR1-specific T cells; Fludarabine; Fludarabine Phosphate; Fludara; Cyclophosphamide; Cytoxan; Neosar; Rituximab; Rituxan; Bendamustine; Bendamustine Hydrochloride; Bendamustine HCL; CEP-18083; SDX-105; Treanda
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ROR1R-CAR-T Cells (Experimental): Peripheral blood mononuclear cells (PBMC) collected via venipuncture and/or steady state leukapheresis at discretion of PI. Participants receive a cycle of lympho-depleting chemotherapy as chosen by treating physician 4 to 5 days before ROR1R-CAR-T cell infusion : Fludarabine, Cyclophosphamide, and Rituximab (FCR), Bendamustine and Rituximab (BR), or Fludarabine, Bendamustine, and Rituximab (FBR).
  Dose Escalation Cohort starting dose level of ROR1R-CAR-T cells/kg: 105 cell/kg infused via central venous catheter or by vein on Day 1.
  Dose Expansion Cohort starting dose level of ROR1R-CAR-T cells/kg: MTD from Dose Escalation Cohort.
  Interventions: Procedure: ROR1R-CAR-T Cell Infusion; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Procedure: ROR1R-CAR-T Cell Infusion — Dose Escalation Cohort starting dose level of ROR1R-CAR-T cells/kg: 105 cell/kg infused via central venous catheter or by vein on Day 1.
  Dose Expansion Cohort starting dose level of ROR1R-CAR-T cells/kg: MTD from Dose Escalation Cohort.
Drug: Fludarabine — FCR Regimen: 25 mg/m2 by vein on Days -5, -4, and -3.
  FBR Regimen: 20 mg/m2 by vein Days -5, -4, and -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — FCR Regimen : 250 mg/m2 by vein on Days -5, -4, and -3.
  Other Names: Cytoxan; Neosar
Drug: Rituximab — FCR and FBR Regimen: 375-500 mg/m2 by vein on Day -5.
  BR Regimen: 375-500 mg/m2 by vein on Day -4.
  Other Names: Rituxan
Drug: Bendamustine — BR Regimen: 70-90 mg/m2 by vein on Days -4 and -3.
  FBR Regimen: 30-50 mg/m2 by vein on Days -5 to -3.
  Other Names: Bendamustine Hydrochloride; Bendamustine HCL; CEP-18083; SDX-105; Treanda

SUMMARY:
Gene transfer is a process in which the DNA (genetic material) of certain cells is changed. In this study, gene transfer will be performed on a type of white blood cell (called T cells) to recognize leukemia cells in the same person the T cells were collected from.

The goal of this clinical research study is to learn if it is safe to give these genetically-changed T cells back to patients with CLL/SLL. Researchers also want to learn if these cells can help to attack CLL/SLL cells.

DETAILED DESCRIPTION:
Standard Blood Draw or Leukapheresis (to collect T cells):

If you are found to be eligible to take part in this study, you will have T cells collected from your blood. This will be done by a standard blood draw or a procedure called leukapheresis. Your doctor will determine which is the best method is to collect your T cells.

If blood is collected through a standard blood draw, blood (less than 7 tablespoons) will be drawn over 1-2 days using one or more needle sticks in your arm.

If you are going to have leukapheresis, you may visit the Apheresis Clinic at MD Anderson. For the leukapheresis procedure, you will need to stay seated in a chair and keep both arms still for about 3 hours. Blood will be drawn from 1 arm, white blood cells will be separated from the rest of the blood cells in the leukapheresis machine, and the red cells, platelets, and plasma (liquid part of the blood) will be returned through your other arm. The leukapheresis procedure may require a total of 4-6 hours each day for up to 2 days.

Your white blood cell sample will be sent to a lab at MD Anderson so the genetically-changed T cells can be grown in the lab.

It will take up to about 4 weeks to change and grow enough genetically-changed T cells. If researchers are unable to create a high enough dose of T cells for you in the lab, you may have more blood collected or you will be taken off study. You may have other treatment for CLL/SLL while you wait for production of the genetically-changed T cells. The study doctor will discuss other possible methods of treatment with you.

Study Groups:

You will be assigned to a level of genetically-changed T cells based on when you join this study. Up to 3 levels of genetically-changed T cells will be tested. Up to 6 participants will be enrolled at each level. The first group of participants will receive the smallest number of T cells. Each new group will receive a higher level than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable level of genetically-changed T cells is found, or the highest level being tested is reached (whichever happens first).

When the highest level is found, an additional 12 patients will receive genetically- changed T cells at that level.

Chemotherapy:

Within 4 or 5 days before you receive your T cell infusion, you will receive 1 of 3 different FDA approved, standard combinations of chemotherapy, chosen by your doctor for you. These combinations are each given over 2-3 days, and must be completed before you receive your T cells. The days before you receive your T cells will be referred to as negative days (for example, 5 days before you receive your T cells will be called Day -5). The drug combinations are known as FCR, FBR, and BR.

If you receive FCR, you will receive fludarabine and cyclophosphamide by vein, both over at least 30 minutes each day on Days -5, -4, and -3. You will also receive rituximab by vein over at least 4 hours on Day -5.

If you receive FBR, you will receive fludarabine and bendamustine by vein, both over at least 30 minutes each day on Days -5, -4, and -3. You will also receive rituximab by vein over at least 4 hours on Day -5.

If you receive BR, you will receive bendamustine by vein over at least 30 minutes each day on Days -4 and -3. You will also receive rituximab by vein on Day -4.

No matter what you receive, you will then rest 2 days in which you receive nothing before your T cell infusion.

T cell Infusion(s):

Before your infusion of genetically-changed T cells, you will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

You will receive your genetically-changed T cells over about 30 minutes on Day 1. During the infusion, your vital signs (including your temperature, heart rate, blood pressure, and breathing rate) will be measured every 15 minutes for the first hour, then every 30 minutes for the second hour, and then about 1 hour after that.

If there are still T cells left over after your infusion, and no intolerable side effects are seen during the first 4 weeks after your infusion, you may receive a second infusion. If you do, you may also receive another course of chemotherapy (as described above).

Study Visits:

About 14 days (+/- 7 days) before receiving your T cell infusion:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test if you can become pregnant.
* Because the gene transfer process uses mouse antibodies, this may cause your body to make human antibodies to the mouse-based antibody. These antibodies are called HAMA. Part of the routine blood sample described above will be used to compare against a sample of your blood collected after the treatment is complete, to check if you developed an immune system reaction against these mouse protein antibodies.
* Blood (about 4 tablespoons) will be drawn for baseline research tests to study how your immune system responds after receiving the T cell infusion.
* If the doctor thinks it is needed, you will have computed tomography (CT) scans, positron emission tomography - CT (PET-CT) scans, and/or a bone marrow biopsy to check the status of the disease.

The following tests and procedures will be performed within 24 hours after your T cell infusion, daily (not including weekends or holidays) for the first week after the infusion, then 1, 2, and 3 weeks (+/-3 days), as well as 1 month (+/- 5 days), and 3, 6, and 12 months (+/- 14 days) after the infusion:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn for routine tests. Part of this blood sample will be used to check for HAMA immune system reactions 1, 2, and 3 weeks, as well as 1, 3, 6, and 12 months after your T cell infusion. If you leave the study early, then your blood will be checked for HAMA at that time.
* Blood (about 4 tablespoons) will be drawn for research tests to study how your immune system is responding to the T cell infusion.
* If your doctor thinks it is needed, you may need CT scans, PET-CT scans, and/or a bone marrow biopsy to check the status of the disease (3, 6, or 12 months after the last T cell infusion only).

Length of Study:

You may receive up to 2 T cell infusions, depending on how many T cells are produced. You will not receive a second T cell infusion if the disease gets worse, you have intolerable side effects, or you have difficulty following the study directions. Your participation on this study will be over when you have completed the study visit at 12 months after the last T cell infusion.

Long-Term Follow-Up:

For safety reasons, the FDA requires that patients who receive infusions of stem cells treated with a gene transfer procedure must have long-term follow-up for at least 15 years after receiving the gene transfer. After you have received an infusion of the T cells you will be asked to sign a separate consent form for a long-term follow-up named "Long-Term Follow-Up Study of Recipients of Gene Transfer Research Protocols" (Protocol 2006-0676).

This is an investigational study. The chemotherapy drugs in this study are commercially available and FDA approved. The gene transfer and infusion with genetically-changed T cells are not commercially available or FDA approved for use in this type of disease. Their use in this study is investigational.

Up to 48 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with B cell CLL/SLL, age </= 85 years old, who have active disease that meets 2008 IWCLL/NCI-WG criteria to initiate treatment.
2. Patients who have failed at least one line of a standard treatment, including bendamustine, fludarabine, ibrutinib, or alemtuzumab and require treatment within 2 years of completion of last treatment regimen or untreated patients with del17p by FISH (high-risk) who do not have an allogeneic stem cell transplant option.
3. At least 21 days from last cytotoxic chemotherapy.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) <2.
5. Adequate hepatic function, defined as substance glutamate pyruvate transaminase (SGPT) <3 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <2 x ULN, or considered not clinically significant by the study doctor or designee.
6. Adequate renal function, defined as serum creatinine <2 x ULN.
7. Able to provide written informed consent, and agree to practicing 2 forms of birth control during the study.
8. Patients must have adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of >40% and adequate pulmonary function as indicated by room air oxygen saturation of >94%.

Exclusion Criteria:

1. Surface ROR1 expression by <5% of CLL cells.
2. Positive beta-HCG in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or lactating females.
3. Patients with known systemic allergy to bovine or murine products.
4. Known positive serology for human immunodeficiency virus (HIV) or human anti-mouse antibody (HAMA).
5. Active, uncontrolled autoimmune phenomenon autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura (AIHA, ITP) requiring steroid therapy.
6. Presence of >/= Grade 3 non-hematologic toxicity common terminology criteria (CTC) version 4 from the previous treatment.
7. Concurrent use of investigational therapeutic agent.
8. Prior allogeneic hematopoietic stem-cell transplantation if evidence of donor chimerism persists. Patients with exclusively autologous hematopoiesis are eligible.
9. Refusal to participate in the long-term follow-up protocol (2006-0676).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ROR1R-CAR-T Cells for Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL) | 4 weeks
  MTD defined as highest dose level in which 6 subjects have been treated with at most 1 subject experiencing ROR1R-CAR-T cell-related dose limiting toxicity (DLT). DLT defined as the following:
  * Common Toxicity Criteria for Adverse Effects (CTCAE) Grade ≥ 3 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to underlying malignancy and occurring within 30 days of study product infusion.
  * CTCAE Grades 3-5 allergic reactions related to study cell infusion.
  * CTCAE Grade ≥ 2 autoimmune reaction related to study product infusion.
  * Treatment-related death within 8 weeks of study product infusion.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PHD, BS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org